CLINICAL TRIAL: NCT03106701
Title: Epicardial Ablation in 500 Consecutive Brugada Syndrome Patients
Brief Title: Epicardial Ablation in Brugada Syndrome. An Extension Study of 500 BrS.Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, Department Director, MD, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCCSDonato
Record Dates: First submitted 2017-03-14; First posted 2017-04-10 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: ECG Brugada Pattern
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation (Experimental): Radiofrequency epicardial ablation
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Epicardial Radiofrequency ablation

SUMMARY:
This study represents an extension of a previous study (NCT02641431) on the acute and long-term benefit of epicardial ablation on elimination of both BrS-ECG pattern and VT/VF inducibility in 500 consecutive BrS patients.

DETAILED DESCRIPTION:
According to previous protocol (NCT02641431), 300 additional consecutive selected patients having an ICD implantation will be enrolled up to a total of 500 BrS patients. Echocardiography with cardiac deformation analysis, three-dimensional color-coded voltage, activation and duration electroanatomical maps before and after ajmaline (1mg/kg in 5 minutes) wiil determine the site and the size of the arrhythmogenic substrate as characterized by abnormally prolonged fragmented ventricular potentials and potential wall motion abnormalities. Primary endpoint will be identification and elimination of this electrophysiological substrate by RF applications leading to ECG pattern normalization and VT/VF non-inducibility before and after ajmaline. Patients will be followed up to 10 years after ablation by sequential 12-lead ECG and Holter recording, Echocardiography, ICD interrogation, VT/VF inducibility patterns before and after ajmaline test.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic BrS patients with typical BrS-related symptoms (cardiac arrest or syncope) or without typical BrS-related symptoms (dizziness, palpitations, presyncope, dyspnea) ICD implantation, spontaneous or ajmaline-induced type 1 Br pattern.

Exclusion Criteria:

* Age < 18 years, prior epicardial ablation, pregnancy, co-morbidities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Type 1 BrS-ECG pattern elimination by epicardial ablation before and after ajmaline test. | 1 day after ablation
  Normalization of ECG pattern after elimination by radio-frequency ablation of all abnormal epicardial potentials
VT/VF inducibility | immediately after mapping and ablation
  Programmed stimulation was achieved at twice the diastolic threshold and randomly performed at RV apex and RV outflow tract using up to 3 drive cycle lengths (from 600 to 350ms) and up to three extrastimuli (S2-S4) delivered from the apex and outflow tract of the right ventricle.
Absence of VT/VF | 1,3,6,12,18,24,36,48,60,72,84,96,108,120 months after ablation
  Absence of VT/VF by ICD interrogation

SECONDARY OUTCOMES:
Absence of Br Pattern and RV mechanical abnormalities using echo and cardiac deformation analysis before and after ajmaline test | 3 months
  Abolition of typical BrS-ECG pattern and RV mechanical abnormalities before and after ajmaline.
Absence of VA episodes at EP study | 3 months
  Non-inducibility of VT/VT at programmed electrophysiological study
Absence of Br Pattern at ajmaline test | 6 months
  Normalization of 12-lead ECG recording and echo parameters at baseline and after ajmaline test
Absence of VA episodes | 6 months
  ICD interrogation
Absence of VA episodes | 12 months
  ICD interrogation and ajmaline test
Absence of Br Pattern at ajmaline test | 12 months
  Normalization of 12-lead ECG recording and echo parameters at baseline and after ajmaline test
Absence of Br Pattern at ajmaline test | 18 months
  Normalization of 12-lead ECG recording at baseline and after ajmaline test
Absence of VA episodes | 24 months
  ICD interrogation
Absence of Br ECG pattern after ajmaline test | 24 months
  Normalization of 12-lead ECG recording at baseline and after ajmaline test
Absence of VA episodes at EP study | 36 months
  ICD interrogation
Absence of Br Pattern at ajmaline test | 36 months
  Normalization of 12-lead ECG recording at baseline and after ajmaline test
Absence of Br Pattern at ajmaline test | 48 months
  Normalization of 12-lead ECG recording at baseline and after ajmaline test
Absence of VA episodes at EP study | 48 months up to 120 months
  ICD interrogation

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — IRCCS Policlinico San Donato, Milan
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ciconte G, Santinelli V, Vicedomini G, Borrelli V, Monasky MM, Micaglio E, Giannelli L, Negro G, Giordano F, Mecarocci V, Mazza BC, Locati E, Anastasia L, Calovic Z, Pappone C. Non-invasive assessment of the arrhythmogenic substrate in Brugada syndrome using signal-averaged electrocardiogram: clinical implications from a prospective clinical trial. Europace. 2019 Dec 1;21(12):1900-1910. doi: 10.1093/europace/euz295. PMID 31647530
- [Derived] Ciconte G, Santinelli V, Brugada J, Vicedomini G, Conti M, Monasky MM, Borrelli V, Castracane W, Aloisio T, Giannelli L, Di Dedda U, Pozzi P, Ranucci M, Pappone C. General Anesthesia Attenuates Brugada Syndrome Phenotype Expression: Clinical Implications From a Prospective Clinical Trial. JACC Clin Electrophysiol. 2018 Apr;4(4):518-530. doi: 10.1016/j.jacep.2017.11.013. Epub 2018 Feb 13. PMID 30067493
- [Derived] Pappone C, Ciconte G, Manguso F, Vicedomini G, Mecarocci V, Conti M, Giannelli L, Pozzi P, Borrelli V, Menicanti L, Calovic Z, Della Ratta G, Brugada J, Santinelli V. Assessing the Malignant Ventricular Arrhythmic Substrate in Patients With Brugada Syndrome. J Am Coll Cardiol. 2018 Apr 17;71(15):1631-1646. doi: 10.1016/j.jacc.2018.02.022. PMID 29650119